CLINICAL TRIAL: NCT01988909
Title: An Open-Label Study to Examine the Safety and Efficacy, of WR 279,396 (Paromomycin + Gentamicin Topical Cream) for the Treatment of Cutaneous Leishmaniasis in France
Brief Title: WR 279,396 for the Treatment of Cutaneous Leishmaniasis
Acronym: PAGELEC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P080705
Record Dates: First submitted 2013-11-14; First posted 2013-11-20 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2017-01

CONDITIONS: Cutaneous Leishmaniasis
Keywords: Cutaneous leishmaniasis; Paromomycin + Gentamicin Topical Cream; Safety; Efficacy
MeSH Terms: conditions — Leishmaniasis, Cutaneous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- WR 279,396 (Experimental): All patients with the same Study drug: WR 279,396 (Topical Paromomycin and Gentamicin Cream)
  Interventions: Drug: WR 279,396

INTERVENTIONS:
Drug: WR 279,396 — Paromomycin + Gentamicin Topical Cream

SUMMARY:
The objectives of the study are to evaluate the safety and efficacy of open label treatment with WR 279,396 (topical paromomycin & gentamicin) in patients with non-complicated, non-severe cutaneous leishmaniasis (CL).

DETAILED DESCRIPTION:
Patients with suspected CL will be screened up to a 14 day period for eligibility including parasitology for confirmation of ulcerative CL. Recruitment will primarily be from patients exposed to leishmaniasis. A target enrollment of 30 patients will receive WR 279,396 (15% paromomycin + 0.5% gentamicin topical cream) once daily for 20 days.

The index lesion and all other ulcerated lesions will be assessed for clinical response by measurement of the length and width of area of ulceration. A lesion will be considered to be completely cured if 100% re-epithelialization is observed. Non-ulcerated lesions will also be measured to monitor the total area of exposure of lesions to study drug and will be evaluated for cure.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for the study, patients must:

1. Be male or females ages 2 to 80 years of age, inclusive.
2. Have non-complicated, non-severe CL.
3. Be able to give written informed consent or by their legal representative.
4. Have a diagnosis of CL in at least one lesion by at least one of the following methods: 1) positive culture for promastigotes; 2) microscopic identification of amastigotes in stained lesion tissue and/or 3) by positive polymerase chain reaction (PCR). Patients who have a prior diagnosis of CL within 30 days of the start of treatment are eligible without a confirmatory test during screening.
5. Have at least one ulcerative lesion ≥ 1 cm and < 5 cm, that meets the criteria for an index lesion.
6. Be willing to forego other forms of treatments for CL including other investigational treatment during the study.
7. In the opinion of the investigator, be capable of understanding (or their legal representative) and complying with the protocol.
8. Expect to be located in the area of the clinical site for at least the duration of the screening, 20-day treatment period, and for the followup visits at Days 28 +/- 2 days, 42 +/- 7 days and 100 +/- 14 days.
9. If female and of child-bearing potential, have a negative serum or urine pregnancy test during screening and agree to use an acceptable method of birth control during the treatment phase and for 1 month after treatment is completed.

Exclusion Criteria:

Also, to be eligible for the study, patients must not:

1. Have a prior diagnosis of leishmaniasis where all lesions had healed.
2. Have only a single lesion whose characteristics include any of the following: verrucous or nodular lesion (non-ulcerative), lesion <1 cm in its greatest diameter, lesion in a location that in the opinion of the Investigator is difficult to maintain application of study drug topically.
3. Have a lesion due to leishmania that involves the mucosa or palate.
4. Have signs and symptoms of disseminated disease.
5. Be a female who is breast-feeding.
6. Have an active malignancy or history of solid, metastatic or hematologic malignancy with the exception of basal or squamous cell carcinoma of the skin that has been removed.
7. Have significant organ abnormality, chronic disease such as diabetes, severe hearing loss, evidence of renal or hepatic dysfunction, myasthenia gravis, parkinsonism, impairment of the eighth cranial nerve or clinically significant levels of creatinine, AST, or ALT in the judgment of the investigator.
8. Have received treatment for leishmaniasis (except mercurochrome or local antiseptics) including any medication with pentavalent antimony including sodium stibogluconate (Pentostam), meglumine antimoniate (Glucantime); amphotericin B (including liposomal amphotericin B and amphotericin B deoxycholate); WR 279,396; or other medications containing paromomycin (administered parenterally or topically) within 56 days of starting study treatments, or methylbenzethonium chloride (MBCL); or local or systemic antibiotics of the following families (penicillin, betalactamics, cyclines, synergistin, macrolides, lincosamides, fusidic acid, mupirocin) within 8 days of starting study treatments.
9. Have history of known or suspected hypersensitivity or idiosyncratic reactions to aminoglycosides.
10. Have any other topical disease/condition which would interfere with the objectives of this study.

Ages: 2 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
final clinical cure rate for the index lesion: initial clinical cure | Day 42 or day 100
  Initial clinical cure: 100% reepithelialization (ie, a 0 x 0 length x width measurement) of the lesion at the nominal Day 42 evaluation, or initial clinical improvement followed >50% reepithelialization by Day 100

SECONDARY OUTCOMES:
final clinical cure rate for the index lesion: Relapse | day 42 or day 100
  Relapse is defined as a 10 percent or greater increase in the area of ulceration of the index lesion or a shift from 100% to < 100% re-epithelialization of the index lesion at nominal Day 100 for those patients that had 100% re-epithelialization of the index lesion at nominal Day 42 or before

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Buffet, MD, PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (2):
- France (2):
  - Groupe Hospitalier Pitié-Salpêtrière, Paris
  - Centre d'investigations cliniques- Hopital Robert Debré, Paris